CLINICAL TRIAL: NCT03561467
Title: Community and Hospital Experiences for Patients Treated by Oral Chemotherapy at the University Hospital of Caen: Analysis of the Process and Its Dysfunctions
Brief Title: Oral Chemotherapy and Quality of Care
Acronym: PARCOURS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Collaborators: MSD France (Industry)
Responsible Party: Sponsor
Other Study IDs: 17-134
Record Dates: First submitted 2018-05-25; First posted 2018-06-19 (Actual); Last update posted 2018-06-19 (Actual); Status verified 2018-05

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Observational — Evaluation of dysfunctions in the continuous city-hospital journey of a patients cohort treated by oral chemotherapy

SUMMARY:
PARCOURS is a non-interventional research study evaluating dysfunctions in the continuous city-hospital journey of a patients cohort treated by oral chemotherapy (60 patients followed for 3 months).

References used are the National Cancer Institute recommendations for the oral chemotherapy treated outpatients.

Parameters found are : information exchanged, ambulatory and hospital monitoring in case of adverse event and adherence to treatment. The study includes also a medico-economic evaluation (hospitalization and transport spending in case of dysfunction in the patient's journey). Deviations will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years old
* Suffering from cancer (hematological malignancies, digestive tumors, thoracic tumors or cutaneous tumors)
* With an oral anticancer chemotherapy initial prescription written by an oncologist or hematologist from the University Hospital of Caen, whatever the place of the drug dispensing (Community pharmacy or hospital pharmacy )

Exclusion Criteria:

- Patient treated by oral anticancer chemotherapy for another pathology

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult outpatients treated by oral chemotherapy for a cancer disease
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2018-03-29 (Actual); Primary Completion 2018-06-29 (Estimated); Study Completion 2018-09-29 (Estimated)

PRIMARY OUTCOMES:
Number of dysfunctions | 3 months
  Number of dysfunctions objectified during the 3-month follow-up period, by sub-processes of the course

SECONDARY OUTCOMES:
Drug adherence | 3 months
  measured by Morisky-Green's questionnaire to the patient
Drug adherence | 3 months
  measured by Data on the refill of prescriptions with the National Health Insurance, and evaluated according to the Drug Possession Ratio
Adverse events | 3 months
  number
Expenses related to the use of unplanned hospital care | 3 months
  Expenses related to the use of unplanned hospital care during the follow-up period: number of oncologist consultations, transport spending, emergency rehospitalizations and additional examinations.
Satisfaction of the patient | At month 3
  RESOCAN questionnaire
Satisfaction of the caregiver | At month 3
  RESOCAN questionnaire
Satisfaction of the local professionals | At month 3
  RESOCAN questionnaire
Quality of life of patients | At month 3
  QLQC 30

CONTACTS AND LOCATIONS:
Locations (1):
- Caen University Hopsital, Caen, France